CLINICAL TRIAL: NCT05984420
Title: Comparative Clinical Trial Between LimpiAD 2.5% Plus Cream, Its Vehicle and a Basic Emollient in Atopic Dermatitis in Paediatric Age
Brief Title: Comparison of LimpiAD Cream 2.5% Plus Versus Its Vehicle and and a Basic Emollient in Patients With Atopic Dermatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aileens Pharma SRL (Industry)
Collaborators: Advice Pharma Group srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LAD-01-21
Record Dates: First submitted 2023-07-25; First posted 2023-08-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis
Keywords: pediatric atopic dermatits; topical medical device; LimpiAD; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Emollients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group LimpiAD (Experimental): LimpiAD 2,5% plus cream to be applied twice a day (morning and evening) for 8 weeks
  Interventions: Device: LimpiAD 2,5% plus cream
- Control group Vehicle of LimpiAD (Active Comparator): Vehicle of LimpiAD 2,5% plus cream to be applied twice a day (morning and evening) for 8 weeks.
  Interventions: Other: Vehicle
- Control group Emollient (Active Comparator): Emollient standard cream to be applied twice a day (morning and evening) for 8 weeks.
  Interventions: Other: Emollient

INTERVENTIONS:
Device: LimpiAD 2,5% plus cream — A topical formulation that contains Hyaluronic Acid conjugated with a bacterial wall fragment of Cutibacterium species (HAc-40) and an emollient base. LimpiAD exerts its post-biotic action through the seizure/ trapping and inactivation of catabolites and / or toxins produced by S. aureus as well as protecting the hydrolipidic film, especially in case of dryness, itching, and, in conditions of altered microbiome
  Arms: Treatment group LimpiAD
Other: Vehicle — Vehicle of LimpiAD 2.5 % plus cream which has the qualities of an emollient technically enriched with active ingredients known for their use in AD ("plus" emollient) - having the same ingredients of LimpiAD 2.5% Plus but without the HAc-40 component.
  Arms: Control group Vehicle of LimpiAD
Other: Emollient — Standard emollient used as neutral control, having only a moisturizing and skin barrier action, which represents the basic standard treatment (basic therapy) of atopic dermatitis according to the European Guidelines.
  Arms: Control group Emollient

SUMMARY:
The purpose of this clinical trial is to assess the efficacy and tolerability of LimpiAD, a medical device in the formulation of a 2.5% Plus cream, versus the Vehicle of LimpiAD 2,5% Plus cream, and versus a basic emollient in subjects with mild to moderate Atopic Dermatitis.

DETAILED DESCRIPTION:
The objective of this clinical trial is to assess the efficacy and tolerability of LimpiAD, a medical device in the formulation of 2.5% Plus cream, versus the Vehicle of LimpiAD 2,5% Plus cream , and versus a basic emollient in subjects with mild to moderate Atopic Dermatitis.

STUDY DESIGN A controlled, 3-arms randomized, double-blind, multicentre clinical trial within subjects, stratified and balanced based on severity of the Atopic Dermatitis (AD) between LimpiAD 2.5% Plus cream, the Vehicle of LimpiAD 2.5% Plus cream and a basic standard treatment (basic therapy) of AD according to European Guidelines in pediatric subjects with mild to moderate AD.

SAMPLE SIZE Two hundred (200) subjects with Atopic Dermatitis, of whom at least 50 cases with mild severity Atopic Dermatitis (defined by EASI = Eczema Area and Severity Index = 1.0-7.0 and IGA= Investigator's Global Assessment =2) and 50 cases with moderate severity Atopic Dermatitis (defined by EASI 7.1-21.0 and IGA=3).

TREATMENT SCHEDULE AND METHODS Treatment with the investigational product or the control products will occur twice daily (morning and evening) for 8 weeks after cleansing of the treatment area. After the 8 weeks treatment period, the study subjects will undergo a follow-up visit after 12 weeks following the baseline visit (4 weeks after treatment completion).

Clinical assessments will be performed at baseline (T0), and after 2, 4, 8 and 12 weeks (T2, T4, T8 and T12) by means of a daily diary as a reminder.

Primary endpoint: statistically significant improvement of the EASI between T0 and T8 (p<0.05) in the treatment arm (LimpiAD 2.5% Plus cream ) as compared to the Vehicle of LimpiAD 2.5% Plus cream.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes, between 6 months and 16 years of age, Caucasian, in good health, whose parents/tutors provided a written and signed informed consent for participation in the study shall be enrolled. In particular, as regards parents/tutors:

  * Both parents/tutors, in case of joint custody, must provide a written and signed informed consent for the participation of the child in the study according to the instructions provided by the investigators;
  * They must accept to bring the child to the clinical trial facility on predefined visit days according to the instructions provided by the investigators;
  * They must be willing and be able to follow the trial requirements provided by the investigators.

The inclusion criteria provide that:

* Symptoms and signs compatible with a clinical diagnosis of Atopic Dermatitis should be present upon enrollment;
* The clinical severity of AD should correspond to an EASI ranging between 1.0 and 21.0 and an IGA equal to 2 or 3;
* Pruritus severity assessed by means of VAS scale ≥ 4 cm should be referred to the part of the body to be treated, as a requirement for inclusion in the study;
* The clinical assessment should envisage for the patient the indication of a moisturizing/emollient treatment as single therapy for AD (in accordance with European Guidelines on AD treatment).

Exclusion Criteria:

The following items are to be considered as exclusion criteria:

* The application of cortisone-based products on the skin to be treated in the 2 weeks prior to treatment;
* Ongoing use at baseline of antibiotics and systemic anti-inflammatory drugs for AD in the 2 weeks preceding treatment and during the study (paracetamol is allowed at dosages and indications recommended for use as an antipyretic and analgesic);
* Baseline treatment with anti-inflammatory drugs, antihistamines, antitussives and/or inhaled steroids in the 2 previous weeks, retinoids and/or immunosupressants in the previous 6 months.
* Use of systemic steroids in the 4 weeks prior to the study.
* Intense and prolonged sun exposure in the 30 days preceding the screening.
* Severe AD (EASI > 21) or mild/moderate AD requiring any local and/or systemic treatment comprised in the prohibited treatments included in the exclusion criteria;
* Hypersensitivity to the study products.
* Acute or chronic skin diseases - except for atopic eczema - which may invalidate clinical assessments or overlap with AD skin picture;
* Systemic diseases which may affect the subject's safety or wellbeing or interfere with skin response.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) | Baseline (T0), 2 weeks (T2), 4 weeks (T4) and 8 weeks (T8)
  The change shall be calculated by comparing the baseline value (T0) with the 2 weeks (T4), 4 weeks (T4) and 8 weeks (T8) values of LimpiAD 2.5% Plus cream versus the Vehicle of LimpiAD 2.5% Plus cream in terms of:
  - score reduction detected (total EASI score)
  INTERPRET EASI: Clear 0; Almost clear 0.1-1.0 ; Mild 1.1-7.0 ; Moderate 7.1-21.0 ; Severe 21.1-50.0; Very severe 50.1-72.0

SECONDARY OUTCOMES:
Change in Investigator Global Assessment (IGA) scale for Atopic Dermatitis | Baseline (T0), 2 weeks (T2), 4 weeks (T4) and 8 weeks (T8)
  The change shall be calculated by comparing the baseline value (T0) of IGA with the 2 weeks (T2), the 4 weeks (T4) and 8 weeks (T8) values in the treatment arm with LimpiAD 2.5% Plus cream as compared to the other 2 arms.
  INTERPRET IGA: 0 - Not affected; 1 - Little affected; 2 - Mild erythema; 3 - Moderate erythema; 4 - Severe Marked erythema
Eczema Area and Severity Index (EASI) Change | Baseline (T0), 2 weeks (T2), 4 weeks (T4) and 8 weeks (T8)
  The change shall be calculated, by comparing the baseline value (T0) with the 2 weeks (T2), 4 weeks (T4) and 8 weeks (T8) values in the treatment arm with LimpiAD 2.5% Plus cream as compared to the other 2 arms in terms of:
  * % of attainment of EASI <1 (corresponding to "healed/almost healed")
  * % of patients reaching a 50% (EASI50), 75% (EASI75), 90% (EASI90) and 100% (EASI100) reduction in the baseline score.
Change in pruritus | Baseline (T0), 4 weeks (T4) and 8 weeks (T8)
  Change in pruritus at the 4 weeks (T4) and 8 weeks (T8). By improvement we mean a Visual Analogue Scale (VAS) reduction below 4 cm, with at least 2-score deviation from baseline (T0), including only the cases with VAS > 5 cm at baseline, in the treatment arm with LimpiAD 2.5% Plus cream as compared to the other 2 treatment arms of the study.
  In the visual analogue scale (VAS), patients are asked to mark on a 10-cm ruler ranging from 0 (no itch) to 10 (worst imaginable itch).
Change in sleep | Baseline (T0), 4 weeks (T4) and 8 weeks (T8)
  Change in sleep at the 4 weeks (T4) and 8 weeks (T8). By improvement we mean a a Visual Analogue Scale (VAS) reduction below 4 cm, with at least 2-score deviation from baseline (T0), including only the cases with VAS > 5 cm at baseline, in the treatment arm with LimpiAD 2.5% Plus cream as compared to the other 2 treatment arms of the study.
  In the visual analogue scale (VAS), patients are asked to mark on a 10-cm ruler ranging from 0 (no disturbance sleep) to 10 (very much disturbed sleep).
Change in extension and signs intensity of the target areas, | Baseline (T0),2 weeks (T2), 4 weeks (T4) and 8 weeks (T8)
  Change in extension and signs intensity of the target areas, assessed as local EASI, by separately considering the skin fold area with respect to the fold-free skin area at 2 weeks (T2), 4 weeks (T4) and 8 weeks (T8) in the treatment arm with LimpiAD 2.5% Plus cream as compared to the other 2 treatment arms of the study.
Children's Dermatology Life Quality Index (CDLQI) questionnaire | Baseline (T0),2 weeks (T2), 4 weeks (T4) and 8 weeks (T8)
  Change in Children's Dermatology Life Quality Index (CDLQI): the change shall be calculated, by comparing the baseline total points (T0) with the corresponding total points at 2 weeks (T2), 4 weeks (T4) and 8 weeks (T8) in the treatment arm with LimpiAD 2.5% Plus cream as compared to the other 2 study treatment arms in terms of:
  -% of achievement of CDLQI <10
  -CDLQI average score reduction
  The CDLQI has 11 questions asking about the impact of a atopic dermatitis on the life of the affected child over the last week.
  Interpretation of QoL: 0-2 = no effect on QoL, 3-7 small effect, 8-13 moderate effect, 14-19 very large effect, 20-33 extremely large effect

CONTACTS AND LOCATIONS:
Overall Officials: Ruggiero Giuseppe, MD, Principal Investigator — ASL Salerno
Locations (5):
- Italy (5):
  - Dr. Chianese Pierluigi, Castellammare di Stabia, Napoli
  - Dr. Carlomagno Francesco, Nola, Napoli
  - Dr. D'Onofrio Antonietta, Pomigliano d'Arco, Napoli
  - Dr. Giuseppe Ruggiero, Battipaglia, Salerno
  - Dr. Occhinegro Aurelio, Salerno

IPD SHARING:
Plan to Share IPD: No